CLINICAL TRIAL: NCT02551185
Title: A Phase 1b Study of the Safety, Pharmacokinetics, and Preliminary Antitumor Activity of ACY 241 in Combination With Paclitaxel in Patients With Advanced Solid Tumors
Brief Title: ACY 241 in Combination With Paclitaxel in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACE-ST-201
Record Dates: First submitted 2015-09-11; First posted 2015-09-16 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — citarinostat

ARMS (1):
- ACY-241 in combination with Paclitaxel (Experimental)
  Interventions: Drug: ACY-241

INTERVENTIONS:
Drug: ACY-241

SUMMARY:
This is a Phase 1b, multicenter, single arm, open label, dose escalation study to determine the MTD and evaluate the safety and preliminary antitumor activity of orally (PO) administered ACY 241 in combination with intravenously (IV) administered paclitaxel in eligible patients with advanced solid tumors.

DETAILED DESCRIPTION:
Patients will receive ACY 241 with dose escalation according to a 3 + 3 design in combination with paclitaxel at the dose and schedule used in clinical practice for the patient population treated in this protocol.

Patients will undergo screening assessments for protocol eligibility within 28 days of study start (Cycle 1 Day 1).

Patients will receive ACY 241 by oral administration once daily (QD) or, if supported by PK and safety data, twice daily on 21 consecutive days of a 28 day treatment cycle. Paclitaxel will be administered to patients at 80 mg/m2 IV over 1 hour on Days 1, 8, and 15 of the 28 day treatment cycle. Patients who experience a DLT or other unacceptable toxicity in Cycle 1 will be removed from study treatment. Patients will receive study treatment until documented progressive disease (PD) or unacceptable toxicity.

Each cohort will consist of at least 3 patients. Patients who withdraw consent in Cycle 1 will be replaced. An assessment of safety will be made by the Safety Review Committee (SRC) before dose escalation. The SRC will be composed of the Study Investigators, the Sponsor's Medical Monitor and Clinical Project Lead, and the Contract Research Organization's Safety Monitor, Project Manager, and Biometrician. Ad hoc members may be invited by the Sponsor as needed.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to understand and voluntarily sign an informed consent form (ICF).
2. Must be ≥ 18 years of age at the time of signing the ICF.
3. Must be able to adhere to the study visit schedule and other protocol requirements.
4. Patients must have a histologically confirmed nonhematological, metastatic or locally advanced, incurable malignancy for which paclitaxel is clinically appropriate. Patients must have received and failed standard treatment for their malignancy; patients for whom no standard treatment is available will also be eligible.
5. Evaluable disease by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
6. Life expectancy > 12 weeks.
7. Must have Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2.
8. Patients with the potential for pregnancy or impregnating their partner must agree to follow acceptable birth control methods to avoid conception. Females of childbearing potential must have a negative pregnancy test. It is not known if the antideacetylase activity of this experimental drug may be harmful to the developing fetus or nursing infant.

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the patient from giving informed consent.
2. Any serious concurrent medical conditions, laboratory abnormality, or psychiatric illness that might make the patient nonevaluable, put the patient's safety at risk, or prevent the patient from following the study requirements.
3. Pregnant or lactating females.
4. Patients with uncontrolled brain metastases.
5. Patients who have had chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) before entering the study or those who have not recovered from AEs to ≤ Grade 1 (except for peripheral neuropathy; see Exclusion Criterion 12) due to agents administered more than 4 weeks earlier.
6. Previous therapy with histone deacetylase (HDAC) inhibitor.
7. Any of the following laboratory abnormalities:

   * ANC < 1,500/µL.
   * Platelet count < 100,000/µL
   * Hematologic growth factors are not allowed at Screening or during the first cycle of treatment.
   * Hemoglobin < 9 g/dL (< 5.5 mmol/L; previous red blood cell [RBC] transfusion is permitted).
   * Creatinine > 1.5 × upper limit of normal (ULN).
   * AST or ALT > 2.5 × ULN. For patients with liver metastasis AST or ALT > 5 × ULN.
   * Serum total bilirubin > 1.5 mg/dL or > 3 × ULN for patients with hereditary benign hyperbilirubinemia
8. Corrected QT interval (QTc) using Fridericia's formula (QTcF) value > 480 msec at Screening; family or personal history of long QTc syndrome or ventricular arrhythmias including ventricular bigeminy at Screening; previous history of drug induced QTc prolongation or the need for treatment with medications known or suspected of producing prolonged QTc intervals on electrocardiogram (ECG).
9. Congestive heart failure (New York Heart Association Class III or IV), myocardial infarction within 12 months before starting study treatment, or unstable or poorly controlled angina pectoris, including Prinzmetal variant angina pectoris.
10. Positive human immunodeficiency virus, hepatitis B virus, and hepatitis C virus infection.
11. Hypersensitivity to taxanes (such as Steven Johnson syndrome). Hypersensitivity, such as rash < Grade 3 that is managed, is allowed.
12. Peripheral neuropathy > Grade 2 despite supportive therapy.
13. Patients who received any of the following within the 14 days before initiating study treatment:

    * Major surgery
    * Radiation therapy
    * Systemic therapy (standard or an investigational or biological anticancer agent)
14. Current enrollment in another clinical study involving treatment and/or is receiving an investigational agent for any reason, or use of any investigational agents within 28 days or 5 half lives (whichever is longer) of initiating study treatment.
15. Incidence of gastrointestinal disease that may significantly alter the absorption of ACY 241.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-12-22 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-04 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLTs) | 12 months
Recommended phase 2 dose and schedule of ACY 241 in combination with paclitaxel on a weekly schedule. | 12 months
Maximum tolerated dose (MTD), if present. | 12 months

SECONDARY OUTCOMES:
Safety profile of ACY 241 administered in combination with paclitaxel. | 12 months
Preliminary antitumor activity of ACY 241 administered in combination with paclitaxel in the patient population. | 12 months

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Pinnacle Oncology Hematology, Scottsdale, Arizona
  - Remove - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - CTRC at The UT Health Science Center at San Antonio, San Antonio, Texas

REFERENCES:
- [Derived] Gordon MS, Shapiro GI, Sarantopoulos J, Juric D, Lu B, Zarotiadou A, Connarn JN, Le Bruchec Y, Dumitru CD, Harvey RD. Phase Ib Study of the Histone Deacetylase 6 Inhibitor Citarinostat in Combination With Paclitaxel in Patients With Advanced Solid Tumors. Front Oncol. 2022 Jan 7;11:786120. doi: 10.3389/fonc.2021.786120. eCollection 2021. PMID 35070991